CLINICAL TRIAL: NCT05074810
Title: A Phase 1/2 Study of Avutometinib (VS-6766) in Combination With Sotorasib With or Without Defactinib in Patients With KRAS G12C Mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase 1/2 Study of Avutometinib (VS-6766) + Sotorasib With or Without Defactinib in KRAS G12C NSCLC Patients
Acronym: RAMP203
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-203
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; KRAS Activating Mutation
Keywords: NSCLC; KRAS G12C
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib; defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- avutometinib (VS-6766)+sotorasib (Experimental): To determine the recommended phase 2 dose (RP2D) for avutometinib (VS 6766) in combination with sotorasib in KRAS G12C inhibitor naïve and exposed patients
  Interventions: Drug: avutometinib and sotorasib
- avutometinib (VS-6766)+sotorasib - KRAS G12C inhibitor naïve (Experimental): To determine the efficacy of the RP2D identified from Part A in KRAS G12C inhibitor naïve patients
  Interventions: Drug: avutometinib and sotorasib
- avutometinib (VS-6766)+sotorasib - KRAS G12C inhibitor exposed (Experimental): To determine the efficacy of the RP2D identified from Part A in KRAS G12C inhibitor exposed patients
  Interventions: Drug: avutometinib and sotorasib
- avutometinib (VS-6766)+sotorasib+defactinib (Experimental): To determine the recommended phase 2 dose (RP2D) for avutometinib (VS-6766) in combination with sotorasib and defactinib in KRAS G12C inhibitor exposed patients
  Interventions: Drug: avutometinib and sotorasib and defactinib
- avutometinib (VS-6766)+sotorasib+defactinib - KRAS G12C inhibitor naive (Experimental): To determine the efficacy of the RP2D identified from Part A in KRAS G12C inhibitor naïve patients
  Interventions: Drug: avutometinib and sotorasib and defactinib
- avutometinib (VS-6766)+sotorasib+defactinib - KRAS G12C inhibitor exposed (Experimental): To determine the efficacy of the RP2D identified from Part A in KRAS G12C inhibitor exposed patients
  Interventions: Drug: avutometinib and sotorasib and defactinib

INTERVENTIONS:
Drug: avutometinib and sotorasib — The RP2D of avutometinib + sotorasib determined in Part A will be used in Part B dose expansion
  Other Names: AMG 510; LUMAKRAS™; VS-6766
  Arms: avutometinib (VS-6766)+sotorasib; avutometinib (VS-6766)+sotorasib - KRAS G12C inhibitor exposed; avutometinib (VS-6766)+sotorasib - KRAS G12C inhibitor naïve
Drug: avutometinib and sotorasib and defactinib — The RP2D of avutometinib + sotorasib + defactinib determined in Part A will be used in Part B dose expansion
  Other Names: AMG 510; LUMAKRAS™; VS-6766; VS-6063
  Arms: avutometinib (VS-6766)+sotorasib+defactinib; avutometinib (VS-6766)+sotorasib+defactinib - KRAS G12C inhibitor exposed; avutometinib (VS-6766)+sotorasib+defactinib - KRAS G12C inhibitor naive

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) in combination with sotorasib with or without defactinib in patients with KRAS G12C Non-Small Cell Lung Cancer (NSCLC) in patients who have been exposed to prior G12C inhibitor and those who have not been exposed to prior G12C inhibitor.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label Phase 1/2 study designed to evaluate safety and tolerability and efficacy of avutometinib (VS-6766) in combination with sotorasib with or without defactinib in patients with KRAS G12C mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Histologic or cytologic evidence of NSCLC
* Known KRAS G12C mutation
* Either exposed or not exposed to a KRAS inhibitor to be included in Part A (avutometinib + sotorasib + defactinib) and not exposed to KRAS inhibitor to be included in Part B (avutometinib + sotorasib + defactinib), Cohort 1
* Received at least 1 dose of a G12C inhibitor to be included in Part B, Cohort 2 (avutometinib + sotorasib + defactinib)
* Must have received appropriate treatment with at least one prior systemic regimen, but no more than 2 prior regimens, for Stage 3B-C or 4 NSCLC
* Measurable disease according to RECIST 1.1
* An Eastern Cooperative Group (ECOG) performance status ≤ 1
* Adequate organ function
* Adequate recovery from toxicities related to prior treatments
* Agreement to use highly effective method of contraceptive

Exclusion Criteria:

* Systemic anti-cancer therapy within 4 weeks of the first dose of study therapy
* History of prior malignancy, with the exception of curatively treated malignancies
* Major surgery within 4 weeks, minor surgery within 2 weeks (excluding placement of vascular access)
* History of treatment with a direct and specific inhibitor of MEK
* Exposure to strong CYP3A4 inhibitors or inducers within 14 days prior to the first dose and during the course of therapy
* Symptomatic brain metastases requiring steroids or other local interventions.
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy
* Known hepatitis B, hepatitis C, or human immunodeficiency virus infection that is active
* Active skin disorder that has required systemic therapy within the past year
* History of rhabdomyolysis
* Concurrent ocular disorders
* Concurrent heart disease or severe obstructive pulmonary disease
* Inability to swallow oral medications
* Female patients that are pregnant or breastfeeding
* Previously treated with sotorasib and were dose reduced due to toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine RP2D for avutometinib in combination with sotorasib and the Alt-RP2D for avutometinib in combination with sotorasib and defactinib | From start of treatment to confirmation of RP2D; 28 days
  Assessment of Dose-limiting toxicities (DLTs)
Part B: To determine the efficacy of the RP2D and/or Alt-RP2D identified from Part A | From start of treatment to confirmation of response; 16 weeks
  Confirmed overall response rate per RECIST 1.1

SECONDARY OUTCOMES:
Frequency and severity adverse events (AEs) and Serious Adverse Events (SAEs) | 24 months
  Count of AE and SAEs by grade, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale
Duration of Response (DOR) | Time from the first documentation of response to first documentation of progressive disease or death due to any cause, greater than or equal to 6 months
  Time of first response to PD as assessed per RECIST 1.1
Disease Control Rate (DCR) | Greater than or equal to 8 weeks
  CR and PR stable disease as assessed per RECIST 1.1
Progression Free Survival (PFS) | 24 months
  From the time of first dose of study intervention to PD or death from any cause
Overall Survival (OS) | Up to 5 years
  From time of first dose of study intervention to death
Plasma Pharmacokinetics (PK) of avutometinib, sotorasib, defactinib and relevant metabolites - Tmax | 10 weeks
  time of Maximum concentration (Tmax)
Plasma Pharmacokinetics (PK) of avutometinib, sotorasib, defactinib and relevant metabolites -AUC | 10 weeks
  Area under plasma Concentration (AUC) 0 to t
Plasma Pharmacokinetics (PK) of avutometinib, sotorasib, defactinib and relevant metabolites half-life | 10 weeks
  concentration Half-life (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: MD Verastem, Study Director — Verastem, Inc.
Locations (35):
- United States (20):
  - Rocky Mountain Cancer Center, LLP, Boulder, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, MedStar Georgetown Cancer Institute,, Washington D.C., District of Columbia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Maryland Oncology & Hematology, P.A., Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A, Woodbury, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Ohio State University Brain and Spine Hospital, Columbus, Ohio
  - Consultants in Medical Oncology & Hematology, Broomall, Pennsylvania
  - Alliance Cancer Specialists,, Horsham, Pennsylvania
  - Texas Oncology, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, Longview, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
- Belgium (2):
  - University Hospital Gent, Ghent
  - CHU de Liège, Liège
- France (3):
  - CHRU of Lille, Lille
  - Hôpital Cochin, Paris
  - Hôpital Foch, Suresnes
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC, Rotterdam
- Spain (5):
  - Hospital Teresa Herrera (C.H.U.A.C), A Coruña
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Universitario Virgen de la Macarena, Seville
- United Kingdom (3):
  - University of Leicester, Leicester
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital, Sutton